CLINICAL TRIAL: NCT07104487
Title: An Exploratory Study of [18F]AlF-NOTA-octreotide PET/MRI in Carotid Artery Disease
Brief Title: [18F]AlF-NOTA-octreotide PET/MRI in Carotid Artery Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S68914; 2024-515636-77 (EudraCT Number)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-10

CONDITIONS: Stroke (CVA) or TIA; Carotid Artery Plaque; Atherosclerosis Cardiovascular Disease; Carotid Arteriosclerosis
Keywords: Internal Carotid Artery; Molecular Imaging; Atherosclerosis; Inflammation; PET/MRI; SST2; [18F]AlF-NOTA-octreotide; Stroke/TIA
MeSH Terms: conditions — Stroke; Carotid Stenosis; Carotid Artery Diseases; Atherosclerosis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Experimental): 5 patients with ≥30% carotid artery stenosis on routine CT angiography (CTA) and a recent ischemic stroke in the supplying carotid artery territory will undergo [18F]AlF-OC PET/MRI at 60, 120 and 180 minutes after tracer injection.
  Interventions: Drug: [18F]AlF-OC
- Arm B (Experimental): 19 patients with ≥30% carotid artery stenosis on routine CTA and a recent ischemic stroke/TIA in the supplying carotid artery territory will undergo [18F]AlF-OC PET/MRI at the timepoint deemed optimal in part A of the study.
  Interventions: Drug: [18F]AlF-OC

INTERVENTIONS:
Drug: [18F]AlF-OC — Participants received a single intravenous (IV) bolus injection of 4 MBq/kg [¹⁸F]AlF-OC (Al¹⁸F-1,4,7-triazacyclononane-1,4,7-triacetate-octreotide), followed by a flush with 0.9% NaCl.

SUMMARY:
This clinical trial aims to evaluate whether [¹⁸F]AlF-OC PET/MRI can characterize and quantify inflammation in carotid atherosclerotic plaques. The study will assess if tracer uptake in culprit and non-culprit carotid arteries, measured by standardized uptake values (SUV), is associated with future cerebrovascular events. Specifically, it will examine whether [¹⁸F]AlF-OC uptake predicts the risk of recurrent ipsilateral TIA, amaurosis fugax, stroke, or other vascular complications.

Participants will undergo [¹⁸F]AlF-OC PET/MRI and will be followed via telephone interviews at 90 days, 1 year, and 3 years after their initial stroke or TIA.

DETAILED DESCRIPTION:
Our study aims to assess the potential of molecular imaging with [18F]AlF-OC PET/MRI to characterize and quantify carotid atherosclerotic disease manifestations in patients with a recent stroke/TIA in the carotid artery territory. Eligible patients should have ≥30% stenosis in the ipsilateral carotid artery, as diagnosed by routine CTA. Additionally, we will evaluate the role of [18F]AlF-OC PET/MRI in risk stratification for recurrent events of patients with carotid artery stenosis and recent TIA/stroke.

This study is a single center study conducted at University Hospitals Leuven in Belgium. In a first part of this study, five patients will undergo serial [18F]AlF-OC PET/MRI at 60, 120 and 180 minutes after injection of 4 MBq/kg [18F]AlF-OC for protocol optimization and methodology refinement. In the second part of this trial, patients will undergo [18F]AlF-OC PET/MRI at the timepoint deemed as optimal based on the findings from the first part. All subjects will be required to undergo a screening and baseline assessment, an imaging visit ([18F]AlF-OC PET/MRI) and three follow-up visits (telephone interview at 90 days, 1 year and 3 years after the initial stroke onset). The primary outcome is the quantification of [18F]AlF-OC uptake in the carotid artery by measures of standardized uptake value (SUV). For every patient, both culprit (recent symptomatic event in ipsilateral carotid artery territory) and non-culprit (recent symptomatic event in the contralateral carotid artery territory) carotid arteries will be assessed. Secondary outcomes include the predictive value of baseline plaque SUV and TBR for the recurrence of ipsilateral TIA, amaurosis fugax and stroke during 3 years follow-up, the recurrence of all stroke/TIA, the occurrence of any vascular complication (stroke/TIA, myocardial infarction, cardiac arrest, hospitalisation for unstable angina or vascular death) and the occurrence of all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged over 18 years.
2. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedure
3. CT angiography imaging at baseline should be available as part of routine care
4. Participant is diagnosed with a recent ischemic stroke or high-risk TIA (ABCD2 ≥ 4) in the carotid artery territory and ≥ 30% carotid artery stenosis. The stroke/TIA has occurred no more than 21 days prior to tracer administration.

Exclusion Criteria:

1. Female who is pregnant or breast-feeding
2. Participants with a cardio-embolic stroke, small vessel stroke or other defined stroke etiology according to the TOAST classification (23)
3. Participant has a previous or ongoing recurrent or chronic disease at high risk to interfere with the performance or evaluation of the trial, according to the judgment of the investigator
4. Participants treated with carotid endarterectomy or carotid artery stenting within the past year
5. Subject has a contra-indication for or cannot tolerate MR scanning
6. Subject has an impaired renal function estimated glomerular filtration rate (eGFR) < 40 ml/min/1.73m² (the last known value may not date from more than 3 months prior to the study PET/MR; if not available a blood analysis may be performed as part of the trial)
7. Concurrent treatment with corticosteroids and/or somatostatin analogues
8. Subject is unwilling or unable to perform all of the study procedures, or is considered unsuitable in any way by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Quantification of ICA [18F]AlF-OC uptake | 1 hour post-injection
  Quantification of [18F]AlF-OC uptake in the culprit and non-culprit carotid artery by measures of standardized uptake value (SUV)

SECONDARY OUTCOMES:
Recurrence of ipsilaterial TIA, stroke or amaurosis fugax | 90 days, 1 year and 3 years after index event
  Recurrence of ipsilateral TIA, amaurosis fugax and stroke during follow-up
Recurrence of all stroke/TIA | 90 days, 1 year and 3 years after the index event
  Recurrence of all stroke/TIA during follow-up
Occurence of major adverse cardiovascular events (MACE) | 90 days, 1 year and 3 years after index event
  Occurence of any vascular complication (stroke/TIA, myocardial infarction, cardiac arrest, hospitalisation for unstable angina or vascular death) during follow-up
Occurence of all-cause mortality | 90 days, 1 year, 3 years after index event
  Occurence of all-cause mortality during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Robin Lemmens, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boeckxstaens L, Pauwels E, Vandecaveye V, Deckers W, Cleeren F, Dekervel J, Vandamme T, Serdons K, Koole M, Bormans G, Laenen A, Clement PM, Geboes K, Van Cutsem E, Nackaerts K, Stroobants S, Verslype C, Van Laere K, Deroose CM. Prospective comparison of [18F]AlF-NOTA-octreotide PET/MRI to [68Ga]Ga-DOTATATE PET/CT in neuroendocrine tumor patients. EJNMMI Res. 2023 Jun 1;13(1):53. doi: 10.1186/s13550-023-01003-3. PMID 37261615
- [Background] Pauwels E, Cleeren F, Tshibangu T, Koole M, Serdons K, Dekervel J, Van Cutsem E, Verslype C, Van Laere K, Bormans G, Deroose CM. [18F]AlF-NOTA-octreotide PET imaging: biodistribution, dosimetry and first comparison with [68Ga]Ga-DOTATATE in neuroendocrine tumour patients. Eur J Nucl Med Mol Imaging. 2020 Dec;47(13):3033-3046. doi: 10.1007/s00259-020-04918-4. Epub 2020 Jul 2. PMID 32617641
- [Background] Maes L, Versweyveld L, Evans NR, McCabe JJ, Kelly P, Van Laere K, Lemmens R. Novel Targets for Molecular Imaging of Inflammatory Processes of Carotid Atherosclerosis: A Systematic Review. Semin Nucl Med. 2024 Sep;54(5):658-673. doi: 10.1053/j.semnuclmed.2023.10.004. Epub 2023 Nov 23. PMID 37996309